CLINICAL TRIAL: NCT06098989
Title: A Prospective Study of REPeat Ablation In Patients With Recurrent PERSistent Atrial Fibrillation: Pulmonary Vein Isolation vs. Adjunct Posterior Wall Isolation (REPAIR PERS-AF Study)
Acronym: REPAIR PERS-AF
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Haukeland University Hospital (Other)
Collaborators: St. Olavs Hospital (Other); University Hospital of North Norway (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 626136
Record Dates: First submitted 2023-10-02; First posted 2023-10-25 (Actual); Last update posted 2023-10-25 (Actual); Status verified 2023-09

CONDITIONS: Atrial Fibrillation, Persistent; Atrial Fibrillation Recurrent
Keywords: Atrial fibrillation; Radiofrequency ablation; Posterior wall isolation; Pulmonary vein isolation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Radiofrequency Ablation

STUDY DESIGN:
Intervention Model Description: Prospective, multi-center, open-labeled, partly randomized study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Normal voltage in LA posterior wall - PVI alone (Active Comparator): Patients with normal LA posterior wall will be assigned directly to arm 1, receiving PVI alone.
  Interventions: Procedure: Radio frequency ablation
- Low voltage in LA posterior wall - PVI alone (Active Comparator): Patients with low voltage/scar on the LA posterior wall will be randomized to arm 2, receiving PVI alone.
  Interventions: Procedure: Radio frequency ablation
- Low voltage in LA posterior wall - PVI + PWI (Active Comparator): Patients with low voltage/scar on the LA posterior wall will be randomized to arm 3, receiving PVI + PWI.
  Interventions: Procedure: Radio frequency ablation

INTERVENTIONS:
Procedure: Radio frequency ablation — Radio frequency ablation

SUMMARY:
This study aims to investigate the best strategy for repeat ablation of recurrent persistent atrial fibrillation (AF) after previous persistent AF ablation involving pulmonary vein isolation (PVI) along. Patients with low voltage areas on the posterer wall will be randomized to PVI alone or the posterer wall isoaltion (PWI) in addition to PVI.

DETAILED DESCRIPTION:
This study aims to find a optmal strategy for repeat ablation for recurrent persistent AF after previous persistent AF ablation involving only PVI. PVI is an evident and well documented target for AF ablation. Many other ablation approaches beyond PVI have been reported. PWI is one of the frequently applied methods. However, this appoach has not been studied in randomized clinical trials for recurrent persistent AF after index procedure, thus evidence is demanded for guidance of clinical practice for AF ablation.

The purpose of this study is to clarify this matter by comparing PVI alone strategy with the approach of PVI plus PWI in patients with recurrent persistent AF after index ablation procedure. Since previous clinical studies have shown better outcomes of ablation among patients with normal left atrium (LA) than those with sick LA, ablation strategies in this study will be selected based on voltage mapping of the LA, avoiding unnecessary ablation applications.

The investigators hypothesize that PVI is good enough for patients with normal LA (normal voltage ≥0.5 mV); Among patients with low voltage/scar (voltage < 0.5 mV), PVI plus PWI is superior to PVI alone.

This study is a prospective, multi-center, open-labeled, partly randomized study. After enrollment, patients will receive a voltage mapping of the LA which is routine for all AF ablation procedures. Based on the mapping results, patients will be stratified into two strata, normal voltage (≥ 0.5 mV) and low voltage (< 0.5 mV) in the LA posterior wall. Patients with normal voltage in the LA posterior wall will be directly assigned to arm 1 receiving PVI alone treatment (avoid unnecessary ablation of healthy myocardium). Patients with low voltage will be 1:1 randomized in arms 2 and 3 receiving either PVI alone or PVI + PWI treatment.

1. Arm 1: Normal voltage in LA posterior wall - PVI alone
2. Arm 2: Low voltage in LA posterior wall - PVI alone
3. Arm 3: Low voltage in LA posterior wall - PVI + PWI

Three Norwegian University Hospitals, including Haukeland University Hospital, Bergen, St. Olavs Hospital, Trondheim, and University Hospital of North Norway, Tromsø, will participate in this study. The study is expected to last 3 years, 24 months for enrollment and each patient will be followed for a period of 12 months.

In order to minimize bias, subjects will be randomized next to the LA mapping. Patients will be analyzed according to their initial randomization, that is intention-to-treat, even if they never start the treatment, or discontinue, or cross over the group.

Patents will be followed in out-patient clinic at 3, 6 and 12 months after the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic patients with persistent AF and indication for repeat ablation
* procedure.
* Patients with recurrent persistent AF (with a duration <3 year, at least one episode longer than 7 days during the last 6 months and have been electrically cardioverted at least once during the last 12 months) after previous catheter ablation.
* Patients with up to two previous catheter ablations for AF are included if the procedures only involved PVI. Previous PVI procedure(s) with both cryoablation and radiofrequency ablation are accepted.
* Patients have taken at least one antiarrhythmic drug.
* Patients are willing to participate in the study and sign the patient information form.
* Age: 18-80 years old.
* Patients must be on continuous anticoagulation with warfarin (INR 2-3) or direct oral anticoagulant for >4 weeks prior to the ablation.

Exclusion Criteria:

* Patients with >2 ablation procedures in the LA for AF or atrial flutter
* Previous ablation procedures for AF involving ablation strategies beyond PVI
* Duration of persistent AF >3 years
* Presence of atrial flutter or atrial tachycardia
* Presence of an intracavitary thrombus
* Uncontrolled heart failure
* Severe valvular disease
* LA diameter > 60 mm
* Structural heart disease involving more than moderate valvular stenosis and/or
* Insufficiencies
* Rheumatic heart disease
* Cardiac surgery for valvopathy or for congenital heart disease
* Patients with contraindications to systemic anticoagulation
* Severe renal dysfunction
* Patients who are or may potentially be pregnant.
* Patient not able to be followed up.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-11-15 (Estimated); Primary Completion 2026-11-15 (Estimated); Study Completion 2026-11-15 (Estimated)

PRIMARY OUTCOMES:
Atrial tachyarrhythmias with duration >30 seconds | 12 months
  Alle episodes of atrial tachyarrhythmia (atrial fibrillation, atrial flutter of atrial tachycardia) with duration >30 seconds recorded 3-months after the ablation procedure will be regarded as recurrence. Blanking period is defined as 3 months.

SECONDARY OUTCOMES:
Complications and adverse events | 12 months
  All periprocedural complications and adverse events during follow-up
Procedure time | During the procedure
  Procedure time will be recorded and reported.
Ablation time | During the procedure
  Ablation time will be recorded and reported.
Fluoroscopy time | During the procedure
  Fluoroscopy time will be recorded and reported.
Quality of life assessment 1 | 12 months
  AF Effect On Quality-Of-Life Questionnaire (AFEQT, scores range 0-100, higher scores mean a worse outcome)
Quality of life assessment 2 | 12 months
  Assessed by Short Form (36) Heath Survey (SF-36, scores range 0-100, higher scores mean a better outcome)
Frequency of atypical atrial flutter | 12 months
  Incidence of atypical atrial flutter will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Jian Chen, MD, PhD, Principal Investigator — Haukeland University Hospital

IPD SHARING:
Plan to Share IPD: No